CLINICAL TRIAL: NCT06242418
Title: Value of CtDNA in Surveillance of Adjuvant Chemosensitivity and Regimen Adjustment in Stage III Colon Cancer: a Phase II Randomized Controlled Trial (REVISE Trial)
Brief Title: CtDNA in Adjuvant Chemotherapy of Stage III Colon Cancer (REVISE Trial)
Acronym: REVISE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Professor, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023#1998
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Colon Cancer
Keywords: colon cancer; ctDNA; adjuvant chemotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — FOLFOXIRI protocol; XELOX

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FOLFOXIRI (Experimental): Eight cycles of FOLFOXIRI: Oxaliplatin 85mg/m2 ivgtt over 2 hours on day 1, Irinotecan 165mg/m2 ivgtt over 90 minutes on day 1, Calcium folinate 400mg/m2 ivgtt over 2 hours on day 1, 5-Fluorouracil 2400mg/m2 civ48h; Each cycle lasts for 2 weeks.
  Interventions: Drug: FOLFOXIRI
- XELOX (Active Comparator): Five cycles of XELOX: Oxaliplatin 130mg/m2 on day 1, Capecitabine 1000mg/m2 bid from day 1 to day 14; Each cycle lasts for 3 weeks.
  Interventions: Drug: XELOX

INTERVENTIONS:
Drug: FOLFOXIRI — Eight cycles of FOLFOXIRI: Oxaliplatin 85mg/m2 ivgtt over 2 hours on day 1, Irinotecan 165mg/m2 ivgtt over 90 minutes on day 1, Calcium folinate 400mg/m2 ivgtt over 2 hours on day 1, 5-Fluorouracil 2400mg/m2 civ48h; Each cycle lasts for 2 weeks.
  Arms: FOLFOXIRI
Drug: XELOX — Five cycles of XELOX: Oxaliplatin 130mg/m2 on day 1, Capecitabine 1000mg/m2 bid from day 1 to day 14; Each cycle lasts for 3 weeks.
  Arms: XELOX

SUMMARY:
Colon cancer is one of the most common malignant tumors with an increasing incidence rate in China. Surgical resection is still the main treatment for colon cancer at present. Radical surgery followed by three/six months chemotherapy is the standard of care for stage III colon cancer; however, patients with different risk factors have different prognosis. The IDEA trial divided stage III colon cancer patients into low-risk (T1-3/N1) and high-risk (T4 or N2) groups, and showed that for some low-risk patients, three months chemotherapy did not decrease survival outcomes, while for some high-risk patients, the recurrence risk was still high even after six months chemotherapy. Therefore, it's worth to explore other risk stratification factors beyond T and N stage for these patients.

Circulating tumor DNA (ctDNA) is derived from cancer cells and can be detected in blood. Literatures have reported that ctDNA can be used for tumor diagnosis, therapeutic monitoring, and prognosis assessment in multiple cancers, including colon cancer. The GERCOR-PRODIGE trial, an accompanying study of IDEA, reported that in the high-risk group of stage III colon cancer, patients with ctDNA-positive and receiving six months chemotherapy had similar prognosis to these with ctDNA-negative and receiving three months chemotherapy; in the low-risk group, patients with ctDNA-negative and receiving three or six months chemotherapy had similar prognosis to patients with ctDNA-positive and receiving 6 months chemotherapy, but patients with ctDNA-positive and receiving three months chemotherapy had the worst prognosis. The results of this trial suggests that ctDNA can be potentially used as a further stratification factor to guide adjuvant chemotherapy for stage III colon cancer.

Several RCTs have shown that double-drug regimens chemotherapy based on oxaliplatin (FOLFOX and XELOX) can improve the prognosis of patients with stage III colon cancer. Therefore, the ESMO, NCCN, and CSCO guidelines recommend FOLFOX or XELOX for stage III colon cancer. The 2-year disease-free survival rate of these patients who received FOLFOX or XELOX chemotherapy was about 80%. It is worth to further explore how to improve the prognosis of these patients. Recently, the triple-drug regimens of oxaliplatin, irinotecan, and fluoropyrimidine (FOLFOXIRI) has been found to be superior to FOLFOX or XELOX for metastatic colorectal cancer in terms of response rate and survival. Currently, research on FOLFOXIRI plus targeted therapy in metastatic colorectal cancer is progressing rapidly, but there is little research on the use of FOLFOXIRI as adjuvant chemotherapy for stage III colon cancer. There is an ongoing international multicenter phase III RCT comparing FOLFOXIRI and FOLFOX6 adjuvant chemotherapy for high-risk stage III colon cancer patients, but it did not further stratify patients based on postoperative ctDNA status, which may result in some patients receiving excessive chemotherapy.

The present study plans to enroll patients with stage III colon cancer with positive ctDNA within 1 month after surgery. These patients will receive 2 cycles of XELOX chemotherapy followed by retesting ctDNA. During the waiting period of the ctDNA results (approximately 3 weeks due to the testing time), all patients will receive another cycle of XELOX chemotherapy. If the ctDNA remains positive, the patients will be randomly assigned to receive 8 cycles of FOLFOXIRI as intensified adjuvant chemotherapy or 5 cycles of XELOX regimen as standard adjuvant chemotherapy. If the ctDNA is negative, the patients will continue to receive 5 cycles of XELOX chemotherapy. Within 3 weeks after the completion or termination of chemotherapy, ctDNA will be retested again. The aims of this study are to explore the value of ctDNA in surveillance of chemosensitivity and to preliminarily evaluate whether the intensified chemotherapy with FOLFOXIRI can increase ctDNA clearance as well as its safety in stage III colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, regardless of gender.
2. Tumor located in the colon (the distance from the lower margin of the tumor to the anus is greater than 12 cm).
3. Radical surgery performed, with pathological stage III (T1-4N1-2M0) (AJCC TNM staging, 8th edition, 2017).
4. No local or distant tumor recurrence was found in imaging examination.
5. Eastern Cooperative Oncology Group (ECOG) performance status: 0-1.
6. adequate organ function: Hemoglobin ≥ 9 g/dL; WBC ≥ 3.5 × 109/ L; Neutrophils ≥ 1.5 × 109/L; Platelets ≥ 100 × 109/L; Creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula); ALT and AST ≤ 2.5 × ULN; Alkaline phosphatase ≤ 2.5 × ULN; Total bilirubin ≤ 1.5 × ULN.
7. No history of allergy to fluoropyrimidines or platinum-based drugs.
8. Voluntarily participating in this study, signing an informed consent form, good compliance, and cooperation with follow-up.

Exclusion Criteria:

1. History of other malignant tumors within the past five years (excluding basal cell carcinoma and/or cervical carcinoma in situ after radical surgery).
2. Patients with BRAF mutation status
3. Patients with microsatellite instability-high (MSI-H) or deficient mismatch repair (dMMR) status
4. Previous chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc., for colon cancer.
5. Patients considering lynch syndrome.
6. Severe cardiovascular or cerebrovascular diseases, liver or kidney dysfunction, severe primary hematological diseases.
7. severe mental disorders
8. Any unstable condition or situation that may harm patient safety or compliance with the study, such as fertility needs, pregnancy, breastfeeding, depression, bipolar disorder, obsessive-compulsive disorder, or schizophrenia.
9. Recently participated in or currently participating in other clinical trials of drugs.
10. Patients deemed unsuitable for participation in this study by the investigator.

Withdrew Criteria

1. Severe adverse reactions to chemotherapy and being unable to continue chemotherapy
2. Metastatic or recurrence disease prior to randomization
3. Refusing further treatment at any time without reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
change in value of ctDNA concentration | six months
  Defined as the change in value of ctDNA measured after 2 cycles of XELOX (ctDNA2) and after the completion or termination of chemotherapy (ctDNA3). △ctDNA= ctDNA3 - ctDNA2.

SECONDARY OUTCOMES:
ctDNA clearance rate | six months
  Defined as the proportion of patients whose ctDNA becomes negative after the completion or termination of chemotherapy to the total patient.
disease-free survival | two years
  The time from randomization to local recurrence, distant metastasis, or death.
metastasis-free survival | two years
  The time from randomization to distant metastasis.
Number of participants with treatment-related adverse events as assessed by CTCAE 5.0. | two years
  Number of participants with treatment-related adverse events as assessed by CTCAE 5.0.
quality of life as assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). | two years
  The EORTC QLQ-C30 consists of 30 items, including 5 functional scales (physical function, role function, cognitive function, emotional function, social function), 3 symptom scales (fatigue, pain, nausea and vomiting), 6 individual measurement items (dysphagia, loss of appetite, sleep disorders, constipation, diarrhea, economic difficulties), and 1 patient self-assessment item (overall health status). Each of the first 28 items score 1 to 4. The higher the score, the worse the quality of life. The last 2 items score 1 to 7. The higher the score, the best the quality of life.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - West China Hospital of Sichuan University, Chengde, Sichuan
  - People's Hospital of Sichuan Province, Chengdu, Sichuan
  - Shang Jin Hospital of West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - The Third People's Hospital of Chengdu, Chengdu, Sichuan
  - West China Tianfu Hospital, Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yunnan Cancer Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
Researchers are encouraged to apply for the full study protocol, study data, and analytic code upon reasonable request by contacting the primary investigator (Ziqiang Wang).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

REFERENCES:
- [Derived] Zhou J, Huang J, Zhou Z, Fan R, Deng X, Qiu M, Wu Q, Wang Z. Value of ctDNA in surveillance of adjuvant chemosensitivity and regimen adjustment in stage III colon cancer: a protocol for phase II multicentre randomised controlled trial (REVISE trial). BMJ Open. 2025 Jan 2;15(1):e090394. doi: 10.1136/bmjopen-2024-090394. PMID 39753246